CLINICAL TRIAL: NCT02106039
Title: Concurrent Tuberculosis and Diabetes: Clinical Monitoring, and Microbiological and Immunological Effects of Diabetes During Tuberculosis Treatment
Brief Title: Pulmonary Tuberculosis Patients With Diabetes Mellitus
Acronym: TANDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other); University of Stellenbosch (Other); St George's, University of London (Other); University of Otago (Other); University of Medicine and Pharmacy Craiova (Other); University Medical Center Groningen (Other); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB-201403.01
Record Dates: First submitted 2014-03-19; First posted 2014-04-07 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus; Pulmonary Tuberculosis
Keywords: diabetes mellitus; tuberculosis; management; randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus; Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive monitoring (Experimental): more intensive monitoring strategy of blood glucose and clinical review
  Interventions: Procedure: intensive monitoring
- standard monitoring (No Intervention): glucose monitoring followed the prevailing practice at each site

INTERVENTIONS:
Procedure: intensive monitoring
  Arms: intensive monitoring

SUMMARY:
The purpose of this study is to evaluate the effect of enhanced glycemic monitoring of diabetes upon diabetes glycaemic control during tuberculosis treatment in tuberculosis- diabetes patients.

DETAILED DESCRIPTION:
Tight glycemic control may improve tuberculosis (TB) treatment outcome and help reduce symptoms. However, active TB and TB treatment hamper glycemic control. Patients starting TB treatment experience rapid changes in appetite, body composition, and inflammation (which increases insulin resistance); inflammation is a feature of untreated TB and following an increase as a result of initial bacterial killing, inflammation subsides with successful treatment. In addition, TB medication (rifampicin) increases the metabolism of oral anti-diabetic drugs including the widely used sulphonylureas and thiazolidinediones, though a possible interaction with the antidiabetic drug metformin has not been previously examined. Frequent monitoring of blood glucose with adjustments in anti-diabetes medication during the course of TB treatment may therefore be needed. However, frequent monitoring is associated with additional costs, and tools and skills for glucose monitoring and diabetes treatment may be lacking in TB or pulmonary clinics, creating a need to refer patients to other health providers. As such, a less intense schedule, preferably following the established decision points in TB treatment after 2 and 6 months would offer significant advantage. None of these issues have been addressed systematically so far.

ELIGIBILITY:
Inclusion Criteria:

* adult (> 18 years old) diabetes mellitus patients
* diagnosed as having active pulmonary TB
* willing to join the study

Exclusion Criteria:

* under TB treatment more than 72 hours
* steroid-induced or gestational diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Better diabetes control in diabetes patients with tuberculosis under treatment | Up to 6 months during TB treatment
  Diabetes control is determined by HbA1c level (unit: %) which will be measured at month 3 and 6 of TB treatment.

SECONDARY OUTCOMES:
Cost-effectiveness of different strategies for diabetes management during TB treatment | Up to 6 months
  Cost analysis will include all cost for lab analysis, transportation for follow up visit, expenses for medications, all complications caused by uncontrolled diabetes (including hospitalization, medications for co morbidities)
Measurement of long-term requirements for diabetes management in TB patients diagnosed with diabetes after TB treatment completed | 12 months after completing TB treatment
  Clinical characteristics (i.e. blood pressure, glucose control, kidney function, quality of life (QoL) of diabetes mellitus patients with TB after completing TB treatment will be measured and will be compared between both groups.
Association between glycemic control and clinical-microbiological response to TB treatment | up to 6 months
  Association between glycemic control and clinical response to TB treatment will be determined by measuring: increasing of body weight, symptoms relieve, treatment outcome (cured, completed, failure and default), and will be compared between groups.
  Association between glycemic control and microbiological response to TB treatment will be determined by measuring sputum conversion time (time to negative culture), and will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Dockrell, Prof, Principal Investigator — London School of Hygiene and Tropical Medicine; Reinout van Crevel, MD, PhD, Study Director — Radboud Universisty Nijmegen Medical Center
Locations (3):
- Faculty of Medicine, Universitas Padjadjaran, Bandung, West Java, Indonesia
- Universidad Peruana Cayetano Heredia, Lima, San Martin de Porres, Peru
- University of Medicine and Pharmacy Craiova, Bucharest, Romania

REFERENCES:
- [Background] Baker MA, Harries AD, Jeon CY, Hart JE, Kapur A, Lonnroth K, Ottmani SE, Goonesekera SD, Murray MB. The impact of diabetes on tuberculosis treatment outcomes: a systematic review. BMC Med. 2011 Jul 1;9:81. doi: 10.1186/1741-7015-9-81. PMID 21722362
- [Background] Ruslami R, Aarnoutse RE, Alisjahbana B, van der Ven AJ, van Crevel R. Implications of the global increase of diabetes for tuberculosis control and patient care. Trop Med Int Health. 2010 Nov;15(11):1289-99. doi: 10.1111/j.1365-3156.2010.02625.x. PMID 20955495
- [Background] Bidstrup TB, Stilling N, Damkier P, Scharling B, Thomsen MS, Brosen K. Rifampicin seems to act as both an inducer and an inhibitor of the metabolism of repaglinide. Eur J Clin Pharmacol. 2004 Apr;60(2):109-14. doi: 10.1007/s00228-004-0746-z. Epub 2004 Mar 19. PMID 15034704
- [Background] Hatorp V, Hansen KT, Thomsen MS. Influence of drugs interacting with CYP3A4 on the pharmacokinetics, pharmacodynamics, and safety of the prandial glucose regulator repaglinide. J Clin Pharmacol. 2003 Jun;43(6):649-60. PMID 12817528
- [Background] Jaakkola T, Backman JT, Neuvonen M, Laitila J, Neuvonen PJ. Effect of rifampicin on the pharmacokinetics of pioglitazone. Br J Clin Pharmacol. 2006 Jan;61(1):70-8. doi: 10.1111/j.1365-2125.2005.02515.x. PMID 16390353
- [Background] Niemi M, Backman JT, Neuvonen M, Neuvonen PJ. Effect of rifampicin on the pharmacokinetics and pharmacodynamics of nateglinide in healthy subjects. Br J Clin Pharmacol. 2003 Oct;56(4):427-32. doi: 10.1046/j.1365-2125.2003.01884.x. PMID 12968988
- [Background] Niemi M, Backman JT, Neuvonen M, Neuvonen PJ, Kivisto KT. Rifampin decreases the plasma concentrations and effects of repaglinide. Clin Pharmacol Ther. 2000 Nov;68(5):495-500. doi: 10.1067/mcp.2000.111183. PMID 11103752
- [Background] Niemi M, Backman JT, Neuvonen M, Neuvonen PJ, Kivisto KT. Effects of rifampin on the pharmacokinetics and pharmacodynamics of glyburide and glipizide. Clin Pharmacol Ther. 2001 Jun;69(6):400-6. doi: 10.1067/mcp.2001.115822. PMID 11406737
- [Background] Niemi M, Kivisto KT, Backman JT, Neuvonen PJ. Effect of rifampicin on the pharmacokinetics and pharmacodynamics of glimepiride. Br J Clin Pharmacol. 2000 Dec;50(6):591-5. doi: 10.1046/j.1365-2125.2000.00295.x. PMID 11136298
- [Background] Park JY, Kim KA, Kang MH, Kim SL, Shin JG. Effect of rifampin on the pharmacokinetics of rosiglitazone in healthy subjects. Clin Pharmacol Ther. 2004 Mar;75(3):157-62. doi: 10.1016/j.clpt.2003.10.003. PMID 15001966
- [Background] Park JY, Kim KA, Park PW, Park CW, Shin JG. Effect of rifampin on the pharmacokinetics and pharmacodynamics of gliclazide. Clin Pharmacol Ther. 2003 Oct;74(4):334-40. doi: 10.1016/S0009-9236(03)00221-2. PMID 14534520
- [Background] Syvalahti E, Pihlajamaki K, Iisalo E. Effect of tuberculostatic agents on the response of serum growth hormone and immunoreactive insulin to intravenous tolbutamide, and on the half-life of tolbutamide. Int J Clin Pharmacol Biopharm. 1976 Mar;13(2):83-9. PMID 1254383
- [Background] Zilly W, Breimer DD, Richter E. Induction of drug metabolism in man after rifampicin treatment measured by increased hexobarbital and tolbutamide clearance. Eur J Clin Pharmacol. 1975 Dec 19;9(2-3):219-27. doi: 10.1007/BF00614021. PMID 1233266
- See also: official website of TANDEM project — http://tandem-fp7.eu